CLINICAL TRIAL: NCT04420988
Title: Investigational COVID-19 Convalescent Plasma Infusion for Severely or Life-threateningly Ill COVID-19 Patients
Status: No longer available | Type: Expanded Access
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: University Hospital - Newark, NJ (Unknown)
Responsible Party: Principal Investigator, Marc Klapholz, M.D., Chair, Department of Medicine; Chief of Medicine Service, University Hospital, Rutgers, The State University of New Jersey
Other Study IDs: Pro2020000746, Pro2020000911
Record Dates: First submitted 2020-05-06; First posted 2020-06-09 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: COVID-19; SARS-CoV 2; SARS-CoV Infection
Keywords: COVID-19 convalescent plasma; convalescent plasma transfusion
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Expanded Access Types: Individual, Intermediate

INTERVENTIONS:
Biological: COVID-19 Convalescent Plasma — COVID-19 Convalescent Plasma from recovered COVID-19 patients transfusion into severely or life-threateningly ill COVID-19 infected patients

SUMMARY:
This is an expanded access program providing COVID-19 convalescent plasma to patients hospitalized with severely or life-threateningly ill COVID-19.

DETAILED DESCRIPTION:
This expanded access program provides hospitalized patients who are severely or life-threateningly ill with COVID-19 access to investigational COVID-19 convalescent plasma (CCP). A clinical team comprised of Infectious Disease specialists, Pulmonary/Critical Care specialists and Hospitalists identify appropriate patients in accordance with FDA recommendations for patient eligibility and the daily availability of ABO-compatible CCP. CCP is obtained through New York Blood Center and American Red Cross in coordination with the University Hospital Blood Bank. Safety outcomes include monitoring for transfusion-related acute lung injury (TRALI), transfusion-associated circulatory overload (TACO) and any allergic reactions.Patients admitted to our institution prior to the availability of CCP will be separately reviewed.

ELIGIBILITY:
Inclusion Criteria:

1. Laboratory confirmed COVID-19.
2. Severe or life-threatening COVID-19. a) Severe disease is defined as one or more of the following: i) dyspnea, ii) respiratory frequency ≥ 30/min, iii) blood oxygen saturation ≤ 93%, iv) partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300, and/or v) lung infiltrates > 50% within 24 to 48 hours b) Life-threatening disease is defined as one or more of the following: i) respiratory failure, ii) septic shock, and/or iii) multiple organ dysfunction or failure

Exclusion Criteria:

1. Contraindication to transfusion (severe volume overload, history of anaphylaxis to blood products)
2. Severe multi-organ failure and hemodynamic instability requiring high doses of pressor agents
3. Other documented uncontrolled infection
4. Severe DIC needing factor replacement, FFP, cryoprecipitate
5. Acute renal failure requiring dialysis
6. Active intracranial bleeding
7. Clinically significant myocardial ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Marc Klapholz, MD, MBA, Principal Investigator — Rutgers New Jersey Medical School; University Hospital
Locations (2):
- United States (2):
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - University Hospital, Newark, New Jersey

REFERENCES:
- [Background] Casadevall A, Scharff MD. Return to the past: the case for antibody-based therapies in infectious diseases. Clin Infect Dis. 1995 Jul;21(1):150-61. doi: 10.1093/clinids/21.1.150. PMID 7578724
- [Background] Casadevall A, Dadachova E, Pirofski LA. Passive antibody therapy for infectious diseases. Nat Rev Microbiol. 2004 Sep;2(9):695-703. doi: 10.1038/nrmicro974. PMID 15372080
- [Background] Zhang JS, Chen JT, Liu YX, Zhang ZS, Gao H, Liu Y, Wang X, Ning Y, Liu YF, Gao Q, Xu JG, Qin C, Dong XP, Yin WD. A serological survey on neutralizing antibody titer of SARS convalescent sera. J Med Virol. 2005 Oct;77(2):147-50. doi: 10.1002/jmv.20431. PMID 16121363
- [Background] Sahr F, Ansumana R, Massaquoi TA, Idriss BR, Sesay FR, Lamin JM, Baker S, Nicol S, Conton B, Johnson W, Abiri OT, Kargbo O, Kamara P, Goba A, Russell JB, Gevao SM. Evaluation of convalescent whole blood for treating Ebola Virus Disease in Freetown, Sierra Leone. J Infect. 2017 Mar;74(3):302-309. doi: 10.1016/j.jinf.2016.11.009. Epub 2016 Nov 17. PMID 27867062
- [Background] Casadevall A, Pirofski LA. Antibody-mediated regulation of cellular immunity and the inflammatory response. Trends Immunol. 2003 Sep;24(9):474-8. doi: 10.1016/s1471-4906(03)00228-x. No abstract available. PMID 12967670
- [Background] Casadevall A, Scharff MD. Serum therapy revisited: animal models of infection and development of passive antibody therapy. Antimicrob Agents Chemother. 1994 Aug;38(8):1695-702. doi: 10.1128/AAC.38.8.1695. No abstract available. PMID 7985997
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Yeh KM, Chiueh TS, Siu LK, Lin JC, Chan PK, Peng MY, Wan HL, Chen JH, Hu BS, Perng CL, Lu JJ, Chang FY. Experience of using convalescent plasma for severe acute respiratory syndrome among healthcare workers in a Taiwan hospital. J Antimicrob Chemother. 2005 Nov;56(5):919-22. doi: 10.1093/jac/dki346. Epub 2005 Sep 23. PMID 16183666
- [Background] Ko JH, Seok H, Cho SY, Ha YE, Baek JY, Kim SH, Kim YJ, Park JK, Chung CR, Kang ES, Cho D, Muller MA, Drosten C, Kang CI, Chung DR, Song JH, Peck KR. Challenges of convalescent plasma infusion therapy in Middle East respiratory coronavirus infection: a single centre experience. Antivir Ther. 2018;23(7):617-622. doi: 10.3851/IMP3243. Epub 2018 Jun 20. PMID 29923831
- [Background] Arabi YM, Hajeer AH, Luke T, Raviprakash K, Balkhy H, Johani S, Al-Dawood A, Al-Qahtani S, Al-Omari A, Al-Hameed F, Hayden FG, Fowler R, Bouchama A, Shindo N, Al-Khairy K, Carson G, Taha Y, Sadat M, Alahmadi M. Feasibility of Using Convalescent Plasma Immunotherapy for MERS-CoV Infection, Saudi Arabia. Emerg Infect Dis. 2016 Sep;22(9):1554-61. doi: 10.3201/eid2209.151164. PMID 27532807
- [Background] van Erp EA, Luytjes W, Ferwerda G, van Kasteren PB. Fc-Mediated Antibody Effector Functions During Respiratory Syncytial Virus Infection and Disease. Front Immunol. 2019 Mar 22;10:548. doi: 10.3389/fimmu.2019.00548. eCollection 2019. PMID 30967872
- [Background] Wan Y, Shang J, Sun S, Tai W, Chen J, Geng Q, He L, Chen Y, Wu J, Shi Z, Zhou Y, Du L, Li F. Molecular Mechanism for Antibody-Dependent Enhancement of Coronavirus Entry. J Virol. 2020 Feb 14;94(5):e02015-19. doi: 10.1128/JVI.02015-19. Print 2020 Feb 14. PMID 31826992
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Chen L, Xiong J, Bao L, Shi Y. Convalescent plasma as a potential therapy for COVID-19. Lancet Infect Dis. 2020 Apr;20(4):398-400. doi: 10.1016/S1473-3099(20)30141-9. Epub 2020 Feb 27. No abstract available. PMID 32113510
- [Background] Duan K, Liu B, Li C, Zhang H, Yu T, Qu J, Zhou M, Chen L, Meng S, Hu Y, Peng C, Yuan M, Huang J, Wang Z, Yu J, Gao X, Wang D, Yu X, Li L, Zhang J, Wu X, Li B, Xu Y, Chen W, Peng Y, Hu Y, Lin L, Liu X, Huang S, Zhou Z, Zhang L, Wang Y, Zhang Z, Deng K, Xia Z, Gong Q, Zhang W, Zheng X, Liu Y, Yang H, Zhou D, Yu D, Hou J, Shi Z, Chen S, Chen Z, Zhang X, Yang X. Effectiveness of convalescent plasma therapy in severe COVID-19 patients. Proc Natl Acad Sci U S A. 2020 Apr 28;117(17):9490-9496. doi: 10.1073/pnas.2004168117. Epub 2020 Apr 6. PMID 32253318
- [Derived] Klapholz M, Pentakota SR, Zertuche JP, McKenna M, Roque W, Forsberg M, Packer J, Lal DS, Dever L. Matched Cohort Study of Convalescent COVID-19 Plasma Treatment in Severely or Life Threateningly Ill COVID-19 Patients. Open Forum Infect Dis. 2021 Jan 4;8(2):ofab001. doi: 10.1093/ofid/ofab001. eCollection 2021 Feb. PMID 33604400

DOCUMENTS (1):
  • Informed Consent Form (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT04420988/ICF_000.pdf